CLINICAL TRIAL: NCT01762137
Title: LARGE Aneurysm Randomized Trial: Flow Diversion Versus Traditional Endovascular Coiling Therapy
Acronym: LARGE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Rarity of disease and current practice in the field made enrollment challenging.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO18426
Record Dates: First submitted 2012-11-16; First posted 2013-01-07 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Intracranial Aneurysm
Keywords: Aneurysm; Coiling; Flow Diversion
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coiling (Active Comparator): Coiling
  Interventions: Procedure: Coiling
- Flow Diversion (Active Comparator): Flow Diversion
  Interventions: Procedure: Flow Diversion

INTERVENTIONS:
Procedure: Flow Diversion — Endovascular flow diverter placement
  Arms: Flow Diversion
Procedure: Coiling — Endovascular coil placement
  Arms: Coiling

SUMMARY:
In this study, patients with large anterior circulation IAs with neck and fundus morphologies amenable to either traditional endovascular treatments using coils or reconstruction with the flow diversion will be randomly assigned to either treatment technique.

DETAILED DESCRIPTION:
This is a prospective, randomized trial comparing the endovascular coiling (endovascular coiling) versus the flow diversion for large and giant aneurysm treatment. The endovascular coiling used in this study are FDA-approved and in common use at institutions in this country and across the world. The flow diversion devices are FDA-approved for anterior circulation aneurysms >10 mm and are in common use at institutions in this country and across the world. Patients will be enrolled who meet the inclusion criteria and consent to participate. Patients will be randomly assigned by a central web-based system in a 1:1 manner to treatment with either endovascular coiling or flow diversion. Data on each patient will be collected at the time of enrollment and treatment, and at subsequent follow-up visits.

ELIGIBILITY:
Inclusion criteria

1. Age 21 to 75 years, inclusive
2. Patient has a single target IA that: is located in the following regions of the internal carotid artery:

   1. Paraophthalmic (including paraclinoid, ophthalmic and hypophyseal segments)
   2. Cavernous
   3. Petrous
3. has a parent vessel with diameter 2.5-5.0 mm
4. Wide neck aneurysm ≥4 mm.
5. Target IA has size (maximum fundus diameter) 10 mm
6. The operator feels that the aneurysm can be appropriately treated with traditional endovascular techniques (endovascular coil embolization with or without adjunctive devices or parent artery deconstruction) using endovascular coiling or flow diversion devices.
7. Modified Rankin Scale 0-3
8. Signed and dated informed consent

4.2 Exclusion criteria

1. More than one IA requiring treatment in the next 6 months
2. Subarachnoid hemorrhage in the past 60 days
3. Any intracranial hemorrhage in the last 42 days
4. Major surgery (requiring general anesthesia) in the last 42 days
5. Coils in place in the target IA
6. Unstable neurologic deficit (i.e., any rapidly worsening clinical condition in the last 30 days (defined by a change in mRS of 2 or more))
7. Known irreversible bleeding disorder
8. Platelet count < 100 x 103 cells/mm3 or known platelet dysfunction
9. Clinically documented evidence in medical history of adverse reaction or contraindication to medications used in treatment of the aneurysm (i.e. Plavix, heparin, aspirin)
10. Prior stent placement at target site
11. Documented history of dementia
12. Contraindication to CT scan and MRI (ie. contrast allergy, or other condition that prohibits imaging from either CT or MRI)
13. Known allergy to contrast used in angiography that cannot be medically controlled
14. Known severe allergy to platinum or cobalt/chromium alloys
15. Relative contraindication to angiography (e.g., serum creatinine > 2.5 mg/dL)
16. Pregnancy, breast-feeding, or positive pregnancy test [either serum or urine] (Woman of child-bearing potential must have a negative pregnancy test prior to the study procedure.)
17. Evidence of active infection (indicated by fever [at or over 99.9 °F] and/or open draining wound) at the time of randomization
18. Other known conditions of the heart, blood, brain or intracranial vessels that carry a high risk of neurologic events (e.g., severe heart failure, atrial fibrillation, known carotid stenosis)
19. Current use of cocaine or other illicit substance
20. Any comorbid disease or condition expected to compromise survival or ability to complete Follow-up assessments through 180 days
21. Extracranial stenosis greater than 50% in the carotid artery
22. Intracranial stenosis greater than 50% in the treated vessel
23. Based on investigator's judgment, patient does not have the necessary mental capacity to participate or is unwilling or unable to comply with protocol follow up appointment schedule.
24. "Previously randomized into this trial or currently participating in another trial where the data is intended to be used to obtain marketing approval or to broaden an indication, without the approval of the study principal investigator, that may confound the results of this study.

A screen failure log of all cases referred or presented for possible inclusion, but who were not randomized, and the reason(s) for exclusion will be maintained.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-02; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
The primary aim of aneurysm treatment is to achieve occlusion of the IA without morbidity or mortality. | approaximately 180 days after aneurysm treatement procedure
  Greater than 90% angiographic occlusion AND stable (or decreased) aneurysm size on cross sectional imaging (CT or MR) at 180 days post procedure. The primary objective is to show that flow diversion is non-inferior to endovascular coiling with respect to a combined efficacy and safety endpoint.

SECONDARY OUTCOMES:
Incidence of device or procedure related adverse events at 180 days, 1 year and 3 years. | approximately 90 days, 180 days, 1 year, 2 year and 3 year
  a count of the occurrences of device related Adverse Events will be recorded and compared between randomized groups at 90, 180, 1year, 2 year, and 3 year time points.
Subgroup analysis of clinical and angiographic outcomes in aneurysms 10-20 mm and > 2 cm. | approximately 3 years after aneurysm treatment procedure
  A comparison will be made as a subgroup analysis of clinical and angiographic outcomes in aneurysms 10-20 mm and > 2 cm. will be measured based on efficacy (Greater than 90% angiographic occlusion AND stable (or decreased) aneurysm size on cross sectional imaging (CT or MR) at 180 days post procedure) and Safety (Free of any major neurologic event (defined as change in NIHSS from baseline > 4 points) downstream from target aneurysm, or death at 180 days post procedure) within this subgroup of study patients.
Downstream flow related ischemic stroke, parenchymal hemorrhage, subarachnoid hemorrhage, aneurysm rupture or re-treatment of index aneurysm rates at 180 days, one year and 3 years. | approaximately 180 days, 1 year, and 3 years after aneurysm treatement procedure
  A count of occurrences of downstream flow related ischemic stroke, parenchymal hemorrhage, subarachnoid hemorrhage, aneurysm rupture or re-treatment of index aneurysm rates at 180 days, one year and 3 years. will be measured and compared at each time point: 180 days, 1 year, and 3 year between groups
Change in clinical functional outcome at 180 days, 1 year and 3 years post-endovascular treatment procedure, as measured by an increase in the modified Rankin Scale from baseline. | 180 days, 1 year and 3 years post-endovascular treatment procedure
  A comparison between groups will be conducted of change in modified rankin scale. The comparison will be measured by an increase in the modified Rankin Scale from baseline, change in clinical functional outcome at 180 days, 1 year and 3 years post-endovascular treatment procedure, as measured by an increase in the modified Rankin Scale from baseline.
Incidence of worsening of baseline neurological signs/symptoms as measured by NIHSS/ophthalmologist exam related to target intracranial aneurysm (IA) at 180 days. | 180 days
  A count and comparison of the incidence of worsening of baseline neurologic signs/symptoms as measured by national institutes of health stroke scale (NIHSS) or ophthalmological exam related to target IA at 180 days will be made between groups.
Number of inpatient hospital (and re-hospitalized) days (subgrouped >7 days) at 180 days, 1 year and 3 years. | 180 days, 1 year and 3 years.
  A count and comparison of the number of inpatient hospital (and re-hospitalized) days (subgrouped >7 days) at 180 days, 1 year and 3 years will be performed between groups
Packing density as measured by volumetric filling of the aneurysm if aneurysm is coiled. | after initial procedure, day 0
  An analysis of packing density as measured by volumetric filling of the aneurysm if aneurysm is coiled will be performed. The analysis will show within group relationships and possible correlations among coiled patients and other variables.
Device cost of therapy at treatment and any subsequent retreatment. | approximately 6 years after the initial procedure
  Device cost of therapy at treatment and any subsequent retreatment will be counted and compared between groups in the study.
Procedure time, as measured as the time from placement of the treating guide catheter for purposes of aneurysm treatment until guide catheter removal. | approximately 6 years after the initial procedure
  Procedure time, as measured as the time from placement of the treating guide catheter for purposes of aneurysm treatment until guide catheter removal, will be collected, measured and compared between groups in the study.
Subgroup analysis of clinical and angiographic outcomes in aneurysms intradural vs. extradural location | approximately 3 years after aneurysm treatment procedure
  A comparison will be made as a subgroup analysis of clinical and angiographic outcomes in aneurysms of intradural vs. extradural location and will be measured based on efficacy (Greater than 90% angiographic occlusion AND stable (or decreased) aneurysm size on cross sectional imaging (CT or MR) at 180 days post procedure) and Safety (Free of any major neurologic event (defined as change in NIHSS from baseline > 4 points) downstream from target aneurysm, or death at 180 days post procedure) within this subgroup of study patients.
Subgroup analysis of clinical and angiographic outcomes in aneurysms reconstructive vs. deconstructive technique. | approximately 3 years after aneurysm treatment procedure
  A comparison will be made as a subgroup analysis of clinical and angiographic outcomes in aneurysms treated with reconstructive vs. deconstructive technique and will be measured based on efficacy (Greater than 90% angiographic occlusion AND stable (or decreased) aneurysm size on cross sectional imaging (CT or MR) at 180 days post procedure) and Safety (Free of any major neurologic event (defined as change in NIHSS from baseline > 4 points) downstream from target aneurysm, or death at 180 days post procedure) within this subgroup of study patients.

CONTACTS AND LOCATIONS:
Overall Officials: Aquilla Turk, DO, Principal Investigator — Medical University of South Carolina
Locations (1):
- MUSC, Charleston, South Carolina, United States